CLINICAL TRIAL: NCT01947010
Title: Pneumococcal Vaccination of Crohn Patients - A Randomized, Non-blinded Phase 4 Clinical Trial With the Purpose of Investigating the Immune Response Against Two Different Pneumococcal Vaccines in Patients With Crohn's Disease
Brief Title: Pneumococcal Vaccination of Crohn Patients
Acronym: PneuVAC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Hvidovre University Hospital (Other); Herlev Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: BJK001
Record Dates: First submitted 2013-09-09; First posted 2013-09-20 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Crohns Disease
Keywords: antibodies
MeSH Terms: conditions — Crohn Disease | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Crohn's patients treated with Azathioprine (Active Comparator): Vaccination with PPV23 or Vaccination with PCV 13
  Interventions: Biological: Prevenar 13; Biological: Pneumovax
- Crohn's patients treated with Azathioprine and TNFa inhibitors (Active Comparator): Vaccination with PPV23 or Vaccination with PCV 13
  Interventions: Biological: Prevenar 13; Biological: Pneumovax
- Crohn's disease patients without treatment (Active Comparator): Vaccination with PPV23 or Vaccination with PCV 13
  Interventions: Biological: Prevenar 13; Biological: Pneumovax

INTERVENTIONS:
Biological: Prevenar 13
Biological: Pneumovax

SUMMARY:
Inflammatory bowel disease (IBD) are at increased risk of infections. This increased susceptibility to infections is due to the disease itself, but also be-cause many patients with autoimmune conditions are treated with immuno-suppressive drugs, such as azathioprine and or TNF-a inhibitors.

Streptococcus pneumoniae (pneumococcus) is a cause of worldwide morbidity and mortality and one of the most common cause of bacterial meningitis in adults. Infection with pneumococcus can be prevented with vaccination. Two pneumococcal vaccine are used in Denmark, the 23 valent polysaccharide-based vaccine (23PPV) and the 13 valent of conjugate pneumococcal vaccines (PCV13).

In this study the investigators wish to study the effect of pneumococcal vaccination with either PPV23 or PCV13 in IBD patients treated with either TNF-a inhibitors, azathioprine or untreated.

DETAILED DESCRIPTION:
Patients with autoimmune diseases like inflammatory bowel disease (IBD) and rheumatoid arthritis (RA) are at increased risk of infections. This increased susceptibility to infections is due to the disease itself, but also be-cause many patients with autoimmune conditions are treated with immuno-suppressive drugs. Different drugs are well-known suppressors of the immune system: Prednisolone, Azathioprine, Methotrexate (MTX), TNF-a inhibitors, and the newer biological agents such as, e.g., Rituximab (RTX), which is a drug used in the treatment of RA patients often in combination with MTX. The extent of immunosuppression induced by these therapeutic agents seems to depend, to some extent, on pharmacological dose/response relationships and on the combination of drugs, but individual variability plays a major role as well.

Prophylactic measures such as vaccination, quick upstart of antibiotics in case of fever and general information to patients about how to handle fever etc. are important in order to prevent as many cases of serious infections as possible among patients in immunosuppressive treatment.

Streptococcus pneumoniae is a cause of worldwide morbidity and mortality. Pneumococcal vaccines have been available since the early 1980's. The vaccine which has been licensed for immunization of children >2 years and adults is a polysaccharide-based vaccine (23PPV) consisting of capsule parts of the 23 most frequent serotypes of pneumococci. This vaccine elicits in normal immunocompetent persons a high antibody response, which lasts for approximately 10 years. Because the 23PPV is a polysaccharide-based vaccine, it induces a T-cell independent response with no memory and there-fore with no possibility of boosting. In 2001, the first generation of conjugate pneumococcal vaccines (PCV7) was licensed. In the PCV's, the capsule material from the pneumococci has been conjugated to a protein, which means that the vaccines can elicit a T-cell dependent immune response even in infants giving memory response and booster possibility. This vaccine has been licensed for use in children from 0-5 years, but studies suggest that PCV immunization might be useful in other groups of people as well etc. immunodeficient children and adults (especially now where the second-generation vaccines PCV10, PCV13 have been licensed covering more pneumococcal serotypes).

Some studies have shown that patients treated with immunosuppressive drugs cannot mount a sufficient antibody response upon vaccination whereas other studies suggest that these patient groups do respond to conventional vaccination.

It is recommended in the Danish guidelines for pneumococcal vaccination, that elderly patients with chronic diseases and patients with a decreased immune system are vaccinated against pneumococcal diseases. Accordingly, patients with Crohn's disease treated with TNF-a inhibitors are recommended pneumococcal vaccination.

In this study, the investigators aim to carry out an investigation of the response to pneumococcal vaccination in persons with Crohn's disease treated with TNF-a inhibitors and/or azathioprine, in order to determine if there is a place for the usage of conjugate vaccination in these patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease, receive immunosuppressive treatment or no treatment

Exclusion Criteria:

* <18 years of age,
* pregnant,
* anemia,
* previously pneumococcus vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in antibody titers | Day 0, 4 weeks post vaccination, 1 year post vaccination
  The primary outcome is to detect a difference in antibody change between the two vaccines as a consequence of the vaccination

SECONDARY OUTCOMES:
Change in antibody titers as a function of Crohns disease treatment | Day 0, 4 weeks post vaccination, 1 year post vaccination
  The secondary outcome is to detect a difference in antibody change between the two vaccines as a function of the treatment for Crohns disease.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Petersen, MD, Principal Investigator — Hvidovre University Hospital; Ole Ø Thomsen, MD, Principal Investigator — Herlev Hospital
Locations (1):
- Statens Serum Institut, Copenhagen, Denmark

REFERENCES:
- [Derived] Kantso B, Halkjaer SI, Ostergaard Thomsen O, Belard E, Gottschalck IB, Jorgensen CS, Krogfelt KA, Slotved HC, Ingels H, Petersen AM. Persistence of antibodies to pneumococcal conjugate vaccine compared to polysaccharide vaccine in patients with Crohn's disease - one year follow up. Infect Dis (Lond). 2019 Sep;51(9):651-658. doi: 10.1080/23744235.2019.1638519. Epub 2019 Jul 10. PMID 31290715
- [Derived] Kantso B, Halkjaer SI, Thomsen OO, Belard E, Gottschalck IB, Jorgensen CS, Krogfelt KA, Slotved HC, Ingels H, Petersen AM. Immunosuppressive drugs impairs antibody response of the polysaccharide and conjugated pneumococcal vaccines in patients with Crohn's disease. Vaccine. 2015 Oct 5;33(41):5464-5469. doi: 10.1016/j.vaccine.2015.08.011. Epub 2015 Aug 12. PMID 26275480